CLINICAL TRIAL: NCT07354282
Title: Retrospective, Multicenter, Real-world Observational Study of Tivozanib as First-line Treatment for Metastatic Clear Cell Renal Cell Carcinoma.
Brief Title: Real World Evidence of Tivozanib as First-line Treatment for Metastatic Clear Cell Renal Cell Carcinoma
Acronym: SOGUG-TIVOREAL
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SOGUG-2024-IEC(REN)-1
Record Dates: First submitted 2025-09-24; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Cancer Metastatic
Keywords: Tivozanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SOGUG-TIVOREAL study is a retrospective observational study with medications.

This study is based on the retrospective collection of data from patients who have been treated with Tivozanib as first-line therapy between 03/01/2019 and 08/31/2024 for metastatic renal cell carcinoma (mRCC).

ELIGIBILITY:
Inclusion Criteria:

1. - Patients ≥ 18 years old.
2. - Who have signed the informed consent form, except for patients who were deceased at the time of inclusion.
3. - Histological diagnosis of stage IV clear cell renal carcinoma.
4. - Who started treatment with Tivozanib as first-line therapy between March 1, 2019, and August 31, 2024.
5. - Who received treatment at the participating center.

Exclusion Criteria:

1. - Patients previously treated at another center who were later referred to one of the participating centers. In this case, the patient will be included in the center where the treatment was initiated.
2. - Explicit objection by the subject or their legal representative to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study consists of patients diagnosed with metastatic renal cell carcinoma (mRCC) who initiated first-line treatment with Tivozanib between March 1, 2019, and August 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Day 1
  To evaluate the progression-free survival (PFS) in patients with metastatic clear cell renal cell carcinoma (mRCC) from the favorable risk group according to IMDC, treated with Tivozanib monotherapy as first-line therapy.
  The probability of progression-free survival will be described using the Kaplan-Meier method, along with the 95% confidence intervals of the point estimates, as well as the median time of survival from the start of treatment with Tivozanib until tumor progression or death from any cause, whichever occurs first. RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) in favorable risk group | Day 1
  To evaluate the overall survival (OS) of patients with metastatic clear cell renal cell carcinoma (mRCC) from the favorable risk group according to IMDC, treated with Tivozanib monotherapy as first-line therapy.
  The probability of overall survival will be described using the Kaplan-Meier method, along with the 95% confidence intervals of the point estimates, as well as the median survival time from the start of treatment with Tivozanib until death from any cause. RECIST 1.1
Objective response rate (ORR) in favorable risk group | Day 1
  To evaluate the objective response rate (ORR) in patients with metastatic clear cell renal cell carcinoma (mRCC) from the favorable risk group according to IMDC, treated with Tivozanib monotherapy as first-line therapy. ORR is defined as the percentage of patients with tumor size reduction (PR) and/or disappearance (CR) after treatment. RECIST 1.1
Percentage of patients with PR and CR in favorable risk group | Day 1
  To evaluate the percentage of patients with partial response (PR) and complete response (CR) among those with metastatic clear cell renal cell carcinoma (mRCC) from the favorable risk group according to IMDC, treated with Tivozanib monotherapy as first-line therapy. RECIST 1.1
Progression-free survival (PFS) - Intermediate and poor risk group | Day 1
  To evaluate the progression-free survival (PFS) in patients with metastatic clear cell renal cell carcinoma (mRCC) from the intermediate and poor risk groups according to IMDC, treated with Tivozanib monotherapy as first-line therapy.
  The probability of progression-free survival will be described using the Kaplan-Meier method, along with the 95% confidence intervals of the point estimates, as well as the median time of survival from the start of treatment with Tivozanib until tumor progression or death from any cause, whichever occurs first. RECIST 1.1
Overall survival (OS) - Intermediate and poor risk group | Day 1
  To evaluate the overall survival (OS) in patients with metastatic clear cell renal cell carcinoma (mRCC) from the intermediate and poor risk groups according to IMDC, treated with Tivozanib monotherapy as first-line therapy.
  The probability of overall survival will be described using the Kaplan-Meier method, along with the 95% confidence intervals of the point estimates, as well as the median survival time from the start of treatment with Tivozanib until death from any cause. RECIST 1.1
Objective response rate (ORR) in poor and intermediate risk group | Day 1
  To evaluate the objective response rate (ORR) in patients with metastatic clear cell renal cell carcinoma (mRCC) from the intermediate and poor risk groups according to IMDC, treated with Tivozanib monotherapy as first-line therapy. ORR is defined as the percentage of patients with tumor size reduction (PR) and/or disappearance (CR) after treatment. RECIST 1.1
Percentage of patients with PR and CR in intermediate and poor risk group | Day 1
  To evaluate the percentage of patients with partial response (PR) and complete response (CR) among those with metastatic clear cell renal cell carcinoma (mRCC) from the intermediate and poor risk groups according to IMDC, treated with Tivozanib monotherapy as first-line therapy. RECIST 1.1
Toxicity profile of Tivozanib | Day 1
  To evaluate the toxicity profile of Tivozanib in the entire study population during the treatment period with Tivozanib, through the evaluation of tivozanib-related toxicities reported in the patients' medical history

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital Reina Sofia, Córdoba, Andalusia
  - Hospital Virgen de la Victoria, Málaga, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital de Burgos, Burgos, Castille and León
  - Hospital de Leon, León, Castille and León
  - Hospital Vall de Hebron, Barcelona, Catalonia
  - Institut Català d'Oncologia (ICO) de L'Hospitalet de Llobregat, L'Hospitalet de Llobregat, Catalonia
  - Hospital Parc Tauli, Sabadell, Catalonia
  - Hospital Lucus Augusti, Lugo, Galicia
  - Hospital Severo Ochoa, Leganés, Madrid
  - Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Instituto Valenciano de Oncologia (IVO), Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No